CLINICAL TRIAL: NCT04978831
Title: The Effect of Use of Breathing Exercise Device and Reading Aloud on Vital Signs, Fatigue and Pulmonary Function Parameters in Patients With COPD Who Followed Up by Wearable Technology
Brief Title: The Effect of Use of Breathing Exercise Device and Reading Aloud on Vital Signs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gürkan ÖZDEN, Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10368355
Record Dates: First submitted 2021-07-17; First posted 2021-07-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Breath Shortness
Keywords: COPD; Fatigue; Breath exercise; Reading aloud
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Respiratory exercise device group (Experimental)
  Interventions: Device: PEP Device
- Reading aloud group (Experimental)
  Interventions: Other: Reading Aloud
- Control group (No Intervention)

INTERVENTIONS:
Device: PEP Device — The breathing exercise device is a device that simulates pursed-lip breathing by creating positive expiratory pressure (PEP). Before starting to use the device, it will be explained that they need to put the mouthpiece on the device and put the nose clip on their nose, and the participants will be shown how it is done. The device will be used at 5 cmH2O pressure. A single exercise session consists of 3 exercise cycles, and a single exercise cycle consists of 15 breathing-exhalation activities. Participants will complete 3 cycles (a total of 45 inhales and exhales) in a single session. 1 loop lying on the left side, 1 loop lying on the right side, and 1 loop in sitting upright position. Participants held these sessions in the morning, afternoon, and evening. After completing each cycle, the participants will remove their nose clips and cough 2-3 times. Each participant will perform a total of 135 breathing exercises in one day.
  Other Names: Smart Watch
  Arms: Respiratory exercise device group
Other: Reading Aloud — The patients in this group were given a book that they chose from among the book types within the scope of the study, according to their wishes. For the selection of books, opinions were taken from the experts in the education faculty of the same university and it was stated that any book separation was not important. The books that the participants wanted to read were provided by the researcher. They were asked to read this book aloud during the day, sitting upright on a chair or sofa, for 15 minutes, three times a day.
  They were able to stop reading when the participant was tired or felt too short of breath to continue reading.
  Arms: Reading aloud group

SUMMARY:
Purpose of the research; To determine the effects of wearable technology follow-up, breathing exercises with a breathing exercise device and reading aloud on vital signs, fatigue and respiratory function parameters in individuals with COPD. This research will be conducted using a randomized controlled trial model. "Personal Description Form", "COPD and Asthma Fatigue Scale", Visual Analog Scale and pulmonary function tests will be used in data collection.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with COPD for at least 6 months or before
* Not having a respiratory system defect caused by diseases other than COPD
* Not in the GOLD-4 COPD stage
* Being able to read and write Turkish
* Have no problems communicating or speaking
* Being able to use basic information technologies
* Using a smartphone
* Having an active internet connection

Exclusion Criteria:

* Having non-COPD pulmonary problems and diagnosed cardiovascular disease
* Not volunteering to participate in the study
* Having a psychiatric disorder such as schizophrenia or dementia that disrupts the thought process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Parameters | 2 month
  Change in FEV1/FVC ratio will be evaluated with pulmonary function test
Fatigue | 2 month
  The COPD and Asthma Fatigue Scale was developed by Revicki et al in 2010 to reveal the effect of COPD and Asthma on fatigue. The items of the questions in the scale, which consists of 12 questions in total, are graded with a 5-point Likert type as "never", "rarely", "sometimes", "often", "very often". A total of 12 to 60 points is obtained from the scale. A single score is obtained from the scale for the state of fatigue, and there is no evaluation of the sub-dimensions. An increase in this score indicates that the person's fatigue level is high.

CONTACTS AND LOCATIONS:
Locations (1):
- İnönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNamara RJ, Epsley C, Coren E, McKeough ZJ. Singing for adults with chronic obstructive pulmonary disease (COPD). Cochrane Database Syst Rev. 2017 Dec 19;12(12):CD012296. doi: 10.1002/14651858.CD012296.pub2. PMID 29253921
- [Background] Wang YT, Green JR, Nip IS, Kent RD, Kent JF. Breath group analysis for reading and spontaneous speech in healthy adults. Folia Phoniatr Logop. 2010;62(6):297-302. doi: 10.1159/000316976. Epub 2010 Jun 28. PMID 20588052